CLINICAL TRIAL: NCT03897608
Title: Quality of Life in Patients With HCV Related Liver Cirrhosis Before and After Direct Acting Antiviral Drugs
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Hossam eldeen Esmael Zayan, RESIDENT DOCTOR, Assiut University
Other Study IDs: life quality with DAAD
Record Dates: First submitted 2019-03-29; First posted 2019-04-01 (Actual); Last update posted 2020-02-11 (Actual); Status verified 2020-02

CONDITIONS: HCV Related Liver Cirrhosis Direct Acting Antiviral Drugs

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: short form 36 — The Short Form (SF)-36 Health Survey was used to measure HRQL. The SF-36 generates a profile of HRQL outcomes by measuring health across eight different dimensions: physical functioning, role limitation because of physical health, social functioning, vitality, bodily pain, mental health, role limitation because of emotional problems and general health. Responses to each question within a dimension are combined to generate a score from 0to100; where100 indicates "good health"

SUMMARY:
To evaluate the effects of DAAs on HRQL in patients with liver cirrhosis secondary to chronic HCV infection

DETAILED DESCRIPTION:
Hepatitis C has been associated with substantial resource utilization as a result of its effect on the liver as well as other organ systems (the extrahepatic manifestations of HCV). It has been widely reported to have a profound negative impact on patient's health-related quality of life (HRQL).

The reduction of HRQL is probably also due to physical and psychiatric symptoms as a direct consequence of this chronic infection and its sequelae (such as cirrhosis). The chronic inflammation is believed to signal the brain and to give rise to neurovegetative symptoms (e.g. malaise and fatigue) and to amongst others depression and concentration difficulties. Possibly, also the brain itself is infected by HCV . The Egyptian government introduced Sofosbuvir as the first DAAs into Egypt through the government funded National Treatment Program. These agents are highly efficacious with significantly fewer side effects .

To date, there is only one study reported about how Egyptian HCV patients receiving the new DAAs perceive their HRQL. This study is first one to be done in Upper Egypt to assess health-related quality of life of HCV patients receiving direct acting antivirals (DAAs) therapy prior and at the end of therapy

ELIGIBILITY:
Inclusion Criteria:

* Patients with hepatitis C related liver cirrhosis (diagnosed clinically laboratory and by imaging).
* Age 18 years or older
* Eligible for starting DAAs therapy according to Egyptian National Guidelines will be enrolled.
* Follow up of those patients during and after DAAs therapy (clinically ,laboratory,imaging and with a questionnaire ) to determine HRQL.

Exclusion Criteria:

* Any patient with liver cirrhosis secondary to causes other than chronic HCV infection e. g. auto immune liver disease, PBC
* Coinfection with other viruses as HBV, HIV.
* Had significant psychiatric illnesses (diagnosed by psychiatrist)

Ages: 11 Months to 12 Months | Sex: All
Age Groups: Child
Study Population: Patients with hepatitis C related liver cirrhosis being treatedusing the Egyptian National Guidelines will be enrolled. According to the most updated treatment protocol, patients undergo therapy for a relatively short period (3 to6 months).
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2020-02-01 (Estimated); Primary Completion 2020-07-01 (Estimated); Study Completion 2020-09-01 (Estimated)

PRIMARY OUTCOMES:
Quality of Life in patients with HCV related liver cirrhosis before and after Direct Acting Antiviral Drugs | one year
  evaluate the effects of DAAs on HRQL in patients with liver cirrhosis secondary to chronic HCV infection

IPD SHARING:
Plan to Share IPD: Undecided